CLINICAL TRIAL: NCT01459900
Title: Renal Sympathectomy in Treatment Resistant Essential Hypertension, a Sham Controlled Randomized Trial
Acronym: ReSET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Silkeborg (Other); Randers Regional Hospital (Other); Regional Hospital Holstebro (Other); Central Jutland Regional Hospital (Other)
Responsible Party: Principal Investigator, Ole Norling Mathiassen, Dr.med, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-20110071
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: Treatment Resistant Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal artery ablation (Active Comparator): By femoral access, coronary and renal angiography are performed. The patient will be sedated. In case of vessel anatomy allowing renal ablation, the patient will be randomized in the card. lab. In case of randomization to active treatment, renal artery ablation will be carried out straight away.
  Interventions: Procedure: Renal artery ablation
- Sham (Sham Comparator): By femoral access, coronary and renal angiography are performed. The patient will be sedated. In case of vessel anatomy allowing renal ablation, the patient will be randomized in the card. lab. In case of randomization to sham procedure, no renal artery ablation are performed.
  Interventions: Procedure: Renal angiography

INTERVENTIONS:
Procedure: Renal artery ablation — Catheter based renal denervation by applying low power radiofrequency to the renal artery using the Ardian Medtronic Simplicity Catheter, introduced by femoral artery access.
  Arms: Renal artery ablation
Procedure: Renal angiography — Renal angiography by femoral access.
  Arms: Sham

SUMMARY:
The purpose of this double blind, randomized and sham controlled study is to determine whether renal denervation in terms of catheter based ablation in the renal arteries is effective in lowering blood pressure in patients with treatment resistant hypertension. The blood pressure lowering effect will be evaluated by 24 hours ambulatory blood pressure measurement at baseline and after 1, 3 and 6 months of follow up. Secondary end point evaluation concerns hemodynamic measures using echocardiography, applanation tonometry and forearm plethysmography.

ELIGIBILITY:
Inclusion Criteria:

* Systolic daytime ambulatory BP at least 145 mmHg and compliance to a minimum of 3 antihypertensive drugs, including a diuretic, or in case of diuretic intolerance at least 3 nondiuretic antihypertensive drugs.

Exclusion Criteria:

* Pregnancy
* Non compliance
* Heart Failure (NYHA 3-4)
* LV ejection fraction < 50 %
* Renal insufficiency (eGFR<30)
* Unstable coronary heart disease
* Coronary intervention within 6 months
* Myocardial infarction within 6 months
* Claudication
* Orthostatic syncope within 6 months
* Secondary Hypertension
* Permanent atrial fibrillation
* Significant Heart Valve Disease
* Clinically Significant abnormal electrolytes, haemoglobin, Liver enzymes, TSH
* Second and third degree heart block
* Macroscopic haematuria
* Proximal significant coronary stenosis
* Renal artery anatomy not suitable for renal artery ablation (Stenosis, small diameter < 4 mm, length < 2 cm, multiple renal arteries, severe calcifications)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
daytime systolic blood pressure assessed by 24 hours ambulatory BP measurement | 3 months follow up
  Changes in mean daytime systolic BP after 3 months is compared between groups. Also the proportion of responders versus nonresponders after 3 months is compared between groups, responders being defined as A) a minimum decrease in daytime systolic BP of 10 mmHg analysis together with and unchanged/increased number of antihypertensive drugs, or B) a decrease in daytime systolic BP of 0-10 mmHg together with a reduced number of antihypertensive drugs.

SECONDARY OUTCOMES:
ambulatory 24 hours BP measurements | 1, 3 and 6 months
  Systolic, diastolic and mean Blood Pressures at different time points. Daytime and night time BP, dipping status, morning BP surge and BP variation.
Echocardiography | 6 months
  Coronary flow reserve (LAD), Diastolic and Systolic ventricular function. LV hypertrophy.
Biomarkers | 1 months
  Biomarkers concerning renal sodium excretion
Applanation tonometry | 6 months
  Pulse wave velocity, augmentation index, central BP estimates
forearm plethysmography | 6 months
  Forearm minimum vascular resistance

CONTACTS AND LOCATIONS:
Overall Officials: Ole N Mathiassen, MD, PhD, Principal Investigator — Aarhus University Hospital, Dep. Cardiology
Locations (1):
- Skejby Hospital, Aarhus, Aarhus N, Denmark

REFERENCES:
- [Derived] Peters CD, Mathiassen ON, Vase H, Bech Norgaard J, Christensen KL, Schroeder AP, Rickers HJVH, Opstrup UK, Poulsen PL, Langfeldt S, Andersen G, Hansen KW, Botker HE, Engholm M, Bertelsen JB, Pedersen EB, Kaltoft A, Buus NH. The effect of renal denervation on arterial stiffness, central blood pressure and heart rate variability in treatment resistant essential hypertension: a substudy of a randomized sham-controlled double-blinded trial (the ReSET trial). Blood Press. 2017 Dec;26(6):366-380. doi: 10.1080/08037051.2017.1368368. Epub 2017 Aug 23. PMID 28830251